CLINICAL TRIAL: NCT02597504
Title: Development of a Neurocognitive Screening Test
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding.
Sponsor: ImPACT Applications, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: QPR-15-44
Record Dates: First submitted 2015-10-16; First posted 2015-11-05 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Brain Concussion; Mild Cognitive Impairment
MeSH Terms: conditions — Brain Concussion; Cognitive Dysfunction | interventions — penclomedine; Prothrombin Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standardization (Active Comparator): individuals assigned to this group will be healthy volunteers and will take the Quick Test.
  Interventions: Device: Quick Test
- Validity and Reliability (Experimental): Reliability:
  Test-Retest
  Validity:
  Concurrent:Quick Test administered with ImPACT online Discriminant: Concussed patient administered Quick Test Construct: Determine agreement between Quick Test and and paper and pencil test.
  Interventions: Other: Pen and paper neuropsychological test; Device: Quick Test

INTERVENTIONS:
Other: Pen and paper neuropsychological test — Will be administered for Construct Validity to determine agreement with Quick Test
  Arms: Validity and Reliability
Device: Quick Test — Quick Test, computerized test will be administered to all subjects.

SUMMARY:
This research study will evaluate a standalone software application and is designed to standardize and validate new neurocognitive screening testing for children aged 6 through 11, and adolescents and adults ages 12 through 75.

The purpose of this study is to evaluate recently developed computerized tasks sensitive to changes in neurocognitive performance after a concussion. These tests were designed to help measure the effects of concussion on cognitive processes (e.g., memory, attention, brain speed) and visual functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-75 (Adult version), 6-11 (pediatric version)
* Primary English speaking or fluent in English.
* No known special education diagnosis excluding a 504 designation.
* Currently not suffering from a concussion or being treated for a concussion.*
* No known physical or psychological impairment that would affect their ability to perform the test.

Exclusion Criteria:

* Documentation of a known special education diagnosis other than a 504 designation.
* English is not their primary language nor are they proficient in the English language.
* Currently suffering from a concussion or being treated for a concussion.*
* Any known physical or psychological impairment that would affect their ability to perform the test.

  * Note: Unless specifically required by the particular study (i.e., a discriminant validity study differentiating concussed versus non-concussed individuals).

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Reliability will be established through a test-retest to establish results should be stable over time | 12 Months
Validity established through correlation studies with well-known measures of memory and processing speed and ANOVA. | 12 Months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - FastMed Urgent Care, Scottsdale, Arizona
  - University of Arkansas, Fayetteville, Arkansas
  - Head First, Crofton, Maryland
  - Jim Gyurke, Pittsburgh, Pennsylvania